CLINICAL TRIAL: NCT07136415
Title: CELESTE: Comparative Effectiveness Study of behavioraL and Drug-rElated inSomnia Therapies for pEri- and Post-menopausal People
Brief Title: Comparing Digital Therapy, Trazodone, and Daridorexant for Menopause-Related Insomnia Symptoms
Acronym: CELESTE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Pittsburgh (Other); University of Utah (Other); Massachusetts General Hospital (Other); Henry Ford Health System (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Suzanne M. Bertisch, MD, MPH, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P001920
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Menopausal Women; Insomnia
Keywords: menopause; insomnia; cognitive behavioral therapy; trazodone; daridorexant
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Trazodone; daridorexant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cognitive behavioral therapy for insomnia (CBT-i) (Active Comparator): Participants will be asked to take part in the CBT-i program over the course of 6-9 weeks, with the option of revisiting content throughout the study duration (12 months).
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBT-i)
- Trazodone (Active Comparator): Participants will be asked to take trazodone (oral pill administration) for the duration of the study (12 months), with safety monitoring conducted by study staff throughout the study. Dosage adjustments may occur.
  Interventions: Drug: Trazodone
- Daridorexant (Active Comparator): Participants will be asked to take daridorexant (oral pill administration) for the duration of the study (12 months), with safety monitoring conducted by study staff throughout the study.
  Interventions: Drug: Daridorexant

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBT-i) — This is a program called SHUT-i and is composed of six self-guided sessions on a website over 6-9 weeks. Each session will be about 45-60 minutes long. CBT-I involves changing behaviors that cause sleep problems to persist. However, it also includes teaching skills to teach the participant to identify thoughts and feelings that may contribute to sleep problems.
  Arms: Cognitive behavioral therapy for insomnia (CBT-i)
Drug: Trazodone — Trazodone is a heterocyclic medication that is FDA-approved for depression (starting dose 150mg). An estimated 4 in 5 trazodone prescriptions are for insomnia. Low-dose trazodone's frequent off-label use stems from a long-standing perception that trazodone is an effective and safer sleep aid compared to other drugs despite potential risks documented in small studies.
  A starting dosage of 25 mg will be used. After 1 week, patients will be instructed to increase the dose as needed to 50mg if tolerated. A second dose adjustment will be made at 4 weeks. At four weeks, study staff will contact participants and review medication adherence, and a standardized checklist will be used to assess ongoing symptoms and side effects and to consider an increase in dose to 100mg.
  Arms: Trazodone
Drug: Daridorexant — Daridorexant is a DORA drug. Dual orexin receptor antagonists (DORAs) are the newest class of FDA-approved medications for insomnia based on efficacy data from pivotal clinical trials demonstrating their efficacy for sleep onset and maintenance.
  A single dose of 50 mg (1 pill each night within 30 minutes of bedtime) was selected based on better efficacy without evidence of higher risks than the 25mg dose.
  Arms: Daridorexant

SUMMARY:
The goal of this clinical trial is to learn how three current insomnia therapies (trazodone, daridorexant, cognitive behavioral therapy for insomnia) compare with each other in peri- and post-menopausal women. It will also learn about the safety of the treatments. The main questions it aims to answer are:

Which commonly used insomnia therapies are most effective and safe for improving insomnia symptoms in peri- and post-menopausal people?

How well do the treatments work for people from different backgrounds, who are at different stages of menopause, and who have different conditions common during menopause (e.g., sleep apnea, mood disturbance, etc.)?

What medical problems do participants have when using these treatments?

Participants will:

Be asked to take trazodone every night, take daridorexant every night, or participate in an online behavioral program for insomnia, for a total of 12 months.

Participate in a total of one in-person visit and 6 virtual visits (phone calls) over the 12 months.

Wear (and keep) a Fitbit and fill out a daily sleep diary for at least 4 weeks over the 12 months.

Fill out online surveys 5 times over the 12 months.

DETAILED DESCRIPTION:
Insomnia, or trouble sleeping, is common. It affects about 1 in 10 adults. People with insomnia are not happy with how long or how well they sleep. Insomnia has been linked to a higher risk of depression, heart disease, memory problems, and lower quality of life. It can also lead to missing work and having accidents. Sleep problems like insomnia are also common or people going through perimenopause and post-menopause.

CBT-I teaches people to change behaviors and thoughts that make it hard to sleep. Daridorexant is an FDA-approved medicine for insomnia. Trazodone is FDA-approved to treat depression, but many doctors also prescribe it to help with sleep. This is called off-label use, which means it is used for a purpose the FDA has not officially approved. Studies show that trazodone is one of the most common medicines prescribed for insomnia in the United States.

We do not yet know how well CBT-I, trazodone, and daridorexant compare, especially for people in perimenopause and post-menopause. Throughout the duration of the study, the participant will be given one of the three therapies.

This study takes about 12 months to complete for each participant.

The following visits and procedures will happen:

Consent telephone or virtual call

Screening Visit: Baseline surveys, urine pregnancy test, electrocardiogram, height and weight assessment. The 7 days after this visit, the participant will also be asked to wear their Fitbit for 24 hours every day, fill out diaries in the morning and night, and wear a home sleep apnea test for one night.

Randomization Call: The participant will be randomized (like a flip of a coin) to receive one of the three insomnia therapies (CBT-I, trazodone, or daridorexant) a week after their baseline visit.

1-week and 4-weeks Call: Quick phone call with study staff for any study treatment adjustments.

3-Months and 6-Months Call/Visit: Fill out surveys. At 6-months, weight will be measured. The 7 days after these visits, the participant will also be asked to wear their Fitbit for 24 hours every day and fill in a sleep diary in the morning and night.

9-Months Call: Quick phone call with study staff to see if there are any issues.

12-Months Call/Visit: Fill out surveys. The 7 days after these visits, the participant will also be asked to wear their Fitbit for 24 hours every day and fill in a sleep diary in the morning and night. The Fitbit is for the participant to keep and does not have to be returned.

ELIGIBILITY:
Inclusion Criteria:

* In peri- or early menopause, following the STRAW criteria of self-report of irregular menstrual cycle or within 5 years from the last menstrual period. In the absence of a reliable menstrual marker (e.g., hysterectomy; endometrial ablation), participants must be older than 45 years old and report hot flashes
* Insomnia severity index score > 10
* Insomnia started or worsened during peri- or early menopause
* English-speaking

Exclusion Criteria:

* Untreated, previously diagnosed severe sleep apnea (self-report; chart review)
* Untreated, previously diagnosed moderate-severe restless legs syndrome (self-report; chart review)
* Severe daytime sleepiness (Epworth Sleepiness Scale > 15)
* Likelihood of limited benefit (e.g., night shift workers with >1 night shift/week; main sleep period outside of 8pm - 11am)
* Regular use of hypnotics > 2 nights/week
* Limited internet access
* Positive urine pregnancy test at baseline visit
* Prolonged QTc interval (>460 ms) (by study baseline electrocardiogram (EKG) or most recent EKG report in medical record)
* History of uncontrolled hypertension or clinically significant heart disease such as arrhythmias requiring medication, cardiomyopathies, heart failure, clinically significant valvular heart disease, or severe coronary artery disease (unstable angina, myocardial infarction in the prior 6 months)
* Use of antiarrhythmics that prolong QTc interval severely (i.e. amiodarone, sotalol, quinidine, procainamide, dofetilide, and ibutilide).
* Known severe chronic liver disease (e.g. cirrhosis)
* History of hypersomnia, narcolepsy, bipolar disorder or psychosis, severe depression, seizure within the past year, use of opioids/substance abuse disorder, pregnant or lactating, , use of strong CYP3A4 inhibitors , use of moderate or strong CYP3A4 inducers, end-stage renal disease on hemodialysis, known allergy to trazodone or daridorexant (self-report and chart review) or other medical condition that increases risk of participation at a study physician's discretion.
* Use of one of the interventions in the past 6 months
* Severe medical comorbidity (e.g., End Stage Renal Disease, likely hospitalization within next 6 months)
* Other conditions determined by the PI to preclude study participation

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Disturbance T-score | 6 Months
  The primary outcome is PROMIS sleep disturbance, which fulfills the criteria for content validity of a patient-reported outcome with reported relevance, comprehensiveness, ease of use, and treatment responses among people with menopause-related insomnia from diverse geographic locations. Sleep disturbance is one of the most bothersome symptoms of the menopause transition and one of the top reasons health care providers report women seek care.
  The PROMIS sleep disturbance scale will be used and the possible range of raw score is 8-40. A higher score means higher levels of sleep disturbance. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
PROMIS Sleep-related Impairment Score | 6 months
  Validated questionnaire assessing daytime alertness. The PROMIS sleep-related impairment scale will be used and the possible range of raw score is 8-40. A higher score means higher levels of sleep-related impairment.
Sleep latency (average) | 6 months
  Measurement of time it takes to fall asleep after going to rest. This is measured in time units (minutes, hours) by self-report and Fitbit. This will be analyzed as a 7-day average.
Client Satisfaction Measure | 6 months
  This is measured via the Client Satisfaction Questionnaire. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Vasomotor Symptoms | 6 months
  The severity and frequency of vasomotor symptoms assessed via self-report and measured by Likert scale and number of hot flashes per day/night, respectively.
Occurrences of events of special interest and/or adverse events | Throughout the study duration (up to 1 year)
  Occurrence of events of special interest (falls, fall-related injuries, drowsiness, dizziness, headache, nausea, dry mouth, palpitations) will be measured for each arm by self-report or chart review. Occurrence of adverse events will also be assessed by number of participants with treatment-related adverse events as defined by CTCAE v4.0
Number of awakenings | 6 months
  Measure of number of awakenings per night by Fitbit.
Sleep duration | 6 months
  Measured by Fitbit, in hours and minutes.
PROMIS Depression Scale | 6 months
  The PROMIS depression scale will be used and the possible range of raw score is 8-40. A higher score means higher levels of depression symptoms.
PROMIS Anxiety Scale | 6 months
  The PROMIS anxiety scale will be used and the possible range of raw score is 8-40. A higher score means higher levels of anxiety symptoms.
PROMIS Cognitive Function Abilities Scale | 6 months
  The PROMIS cognitive function abilities scale will be used and the possible range of raw score is 4-20. A higher score represents better cognitive function.
PROMIS Anger Scale | 6 months
  The PROMIS anger scale will be used and the possible range of raw score is 5-25. A higher score means higher levels of anger.
PROMISE Global Health Score | 6 months
  The PROMIS global health scale will be used and the possible range of raw score is 8-40. A higher score indicates better physical and mental health.
PROMIS Fatigue Score | 6 months
  The PROMIS fatigue scale will be used and the possible range of raw score is 8-40. A higher score indicates higher levels of fatigue.
PROMIS Interest in Sexual Activity Score | 6 months
  The PROMIS interest in sexual activity scale will be used and the possible range of raw score is 2-10. A higher score indicates greater interest in sexual activity.
PROMIS Satisfaction with Sex Life Score | 6 months
  The PROMIS satisfaction with sex life scale will be used and the possible range of raw score is 4-20. A higher score indicates higher satisfaction with sex life.
Menopause-related Quality of Life | 6 months
  The menopause-related quality of life (MENQOL) scale will be used and the possible range of raw score is 29-232. A higher score indicates higher severity of menopause-related symptoms.
Work Productivity and Activity Impairment | 6 months
  The Work Productivity and Activity Impairment - General Health (WPAI-GH) Questionnaire is a 6-item instrument to measure impairments over the past 7 days in both paid work and unpaid work due to one's health. Higher numbers indicate greater impairment and less productivity. Four main outcomes can be yielded from WPAI and are presented as percentages (0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Bertisch, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No